CLINICAL TRIAL: NCT01399424
Title: Shigella Sonnei OSPC-rDT Conjugate Vaccine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Rachel Schneerson, M.D./National Institute of Child Health and Human Development, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999911214; 11-CH-N214
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-25

CONDITIONS: Shigellosis
Keywords: Shigellosis; Safety and Immunogenicity; Conjugate Vaccine; Shigella; Vaccine
MeSH Terms: conditions — Dysentery, Bacillary

INTERVENTIONS:
Drug: CP — Immunization

SUMMARY:
The active ingredient of this Shigella sonnei O-SP-core conjugate vaccine is a saccharide-protein conjugate composed of a fragment of S. sonnei LPS. The saccharide component consists of an average of 3.5 repeat units of the O-SP plus the core region of the LPS (O-SPC). The O-SPC is covalently bound to the non-toxic recombinant diphtheria toxin mutant (rDT).

The objective of this phase of the study is to determine if this vaccine is safe and can induce IgG antibody type-specific immunity to shigellosis in adults. The overall objective is to determine if this vaccine can elicit higher levels of IgG antibody than the previous experimental vaccines made with the full length O-SP, shown to be > 70% efficacious in greater than or equal to 3 year old children. Higher levels of IgG anti O-SP are expected to induce type specific immunity to shigellosis in younger children.

Sixty 18-49 years-old healthy adults will be recruited in Israel. Volunteers will be vaccinated on a random basis with one i.m. injection of 10 or 25 ug of the investigational conjugate vaccine. Local and systemic reactions will be observed at 30 minutes, and the volunteers will be instructed to take their temperature and examine the injection site for redness and swelling and fill out a questionnaire at 6, hours and daily for 7 days after vaccination. The volunteers will visit the clinic at 24 or 48 hours following the injection and any time they request it. The study will commence with 5 volunteers injected with the 10ug dose to be followed, if no severe adverse reactions occur, by 5 volunteers injected with the 25ug dose. If a severe adverse reaction occurs on 1 of the 5 volunteers in either group, 5 more will be injected with that dose. If there are no severe adverse reactions the study will proceed. If there is one more severe reaction the study will be halted and re-evaluated by the IRB and the FDA.

Vaccine-induced antibodies will be measured at 1 and 6 months after immunization, and compared to those elicited by our previous S. sonnei conjugate vaccines.

There is a body of evidence that a critical level of serum IgG antibody to the O-specific polysaccharide domain of LPS confers type-specific immunity to S. sonnei as well as to other Shigella:

1. Shigellosis is rarely observed in infants up to the age of 4-6 months. The most obvious explanation for this is that maternally-derived serum IgG provides this immunity;
2. There is an age-related development of IgG anti-LPS antibodies that, in many instances, is not induced by the homologous bacteria but by non-pathogenic cross-reacting enteric bacteria;
3. The highest incidence, morbidity, and mortality occur during 6 months to 6 years of age when the maternally-derived serum anti-O-SP has waned and the naturally-derived antibodies have not yet appeared;
4. One injection of a S. sonnei-rEPA conjugate showed significant protection against shigellosis in Israeli Defense Force soldiers. Vaccinees who developed shigellosis showed significantly lower serum IgG responses to the homologous LPS than those did not.The high antibody level induced by the conjugate vaccine indicates the positive correlation between the serum IgG anti-LPS levels and immunity to S. sonnei infection;
5. Following Phase 1 and Phase 2 studies that showed safety and age-related immunogenicity, a double-blinded randomized and vaccine-controlled Phase 3 evaluation of S. sonnei and S. flexneri type 2a O-specific polysaccharide (O-SP) protein conjugates was conducted among 1-4 year-olds in Israel.

For recipients of the S. sonnei conjugate 71.1% efficacy was shown among 3-4 year-old recipients, no efficacy was shown for recipients of S. flexneri 2a. There was no statistically significant efficacy for either vaccine in the 1-3 year-olds. Levels of serum IgG anti-O-SP were elevated according to the vaccine the children received but G.M. levels declined rapidly several months after the last injection. Our interpretation is that the age-related efficacy of the Shigella conjugates was due to the conjugate-induced O-SP antibody levels. Accordingly, we have developed a method to increase the immunogenicity of the conjugates to approach the antibody levels of Israeli soldiers shown to be protected by our S. sonnei O-SP.

Low-molecular-mass O-SP-core (O-SPC) fragments were isolated from S. sonnei LPS, and bound by their reducing ends to the carrier protein. The O-SPC conjugates used oxime linkages between the terminal Kdo residues at the reducing ends of the S. sonnei saccharides and aminooxy linkers bound to the carrier. The coupling reaction was carried out at a neutral pH and room temperature. The carrier protein was a non-toxic recombinant diphtheria toxin mutant. IgG antibody levels induced in young outbred mice by this new S. sonnei O-SPC conjugate were significantly higher then those elicited by the O-SP conjugates.

DETAILED DESCRIPTION:
The active ingredient of this Shigella sonnei O-SP-core conjugate vaccine is a saccharide-protein conjugate composed of a fragment of S. sonnei LPS. The saccharide component consists of an average of 3.5 repeat units of the O-SP plus the core region of the LPS (O-SPC). The O-SPC is covalently bound to the non-toxic recombinant diphtheria toxin mutant (rDT).

The objective of this phase of the study is to determine if this vaccine is safe and can induce IgG antibody type-specific immunity to shigellosis in adults. The overall objective is to determine if this vaccine can elicit higher levels of IgG antibody than the previous experimental vaccines made with the full length O-SP, shown to be > 70% efficacious in greater than or equal to 3 year old children. Higher levels of IgG anti O-SP are expected to induce type specific immunity to shigellosis in younger children.

Sixty 18-49 years-old healthy adults will be recruited in Israel. Volunteers will be vaccinated on a random basis with one i.m. injection of 10 or 25 ug of the investigational conjugate vaccine. Local and systemic reactions will be observed at 30 minutes, and the volunteers will be instructed to take their temperature and examine the injection site for redness and swelling and fill out a questionnaire at 6, hours and daily for 7 days after vaccination. The volunteers will visit the clinic at 24 or 48 hours following the injection and any time they request it. The study will commence with 5 volunteers injected with the 10ug dose to be followed, if no severe adverse reactions occur, by 5 volunteers injected with the 25ug dose. If a severe adverse reaction occurs on 1 of the 5 volunteers in either group, 5 more will be injected with that dose. If there are no severe adverse reactions the study will proceed. If there is one more severe reaction the study will be halted and re-evaluated by the IRB and the FDA.

Vaccine-induced antibodies will be measured at 1 and 6 months after immunization, and compared to those elicited by our previous S. sonnei conjugate vaccines.

There is a body of evidence that a critical level of serum IgG antibody to the O-specific polysaccharide domain of LPS confers type-specific immunity to S. sonnei as well as to other Shigella:

1. Shigellosis is rarely observed in infants up to the age of 4-6 months. The most obvious explanation for this is that maternally-derived serum IgG provides this immunity;
2. There is an age-related development of IgG anti-LPS antibodies that, in many instances, is not induced by the homologous bacteria but by non-pathogenic cross-reacting enteric bacteria;
3. The highest incidence, morbidity, and mortality occur during 6 months to 6 years of age when the maternally-derived serum anti-O-SP has waned and the naturally-derived antibodies have not yet appeared;
4. One injection of a S. sonnei-rEPA conjugate showed significant protection against shigellosis in Israeli Defense Force soldiers. Vaccinees who developed shigellosis showed significantly lower serum IgG responses to the homologous LPS than those did not.The high antibody level induced by the conjugate vaccine indicates the positive correlation between the serum IgG anti-LPS levels and immunity to S. sonnei infection;
5. Following Phase 1 and Phase 2 studies that showed safety and age-related immunogenicity, a double-blinded randomized and vaccine-controlled Phase 3 evaluation of S. sonnei and S. flexneri type 2a O-specific polysaccharide (O-SP) protein conjugates was conducted among 1-4 year-olds in Israel.

For recipients of the S. sonnei conjugate 71.1% efficacy was shown among 3-4 year-old recipients, no efficacy was shown for recipients of S. flexneri 2a. There was no statistically significant efficacy for either vaccine in the 1-3 year-olds. Levels of serum IgG anti-O-SP were elevated according to the vaccine the children received but G.M. levels declined rapidly several months after the last injection. Our interpretation is that the age-related efficacy of the Shigella conjugates was due to the conjugate-induced O-SP antibody levels. Accordingly, we have developed a method to increase the immunogenicity of the conjugates to approach the antibody levels of Israeli soldiers shown to be protected by our S. sonnei O-SP.

Low-molecular-mass O-SP-core (O-SPC) fragments were isolated from S. sonnei LPS, and bound by their reducing ends to the carrier protein. The O-SPC conjugates used oxime linkages between the terminal Kdo residues at the reducing ends of the S. sonnei saccharides and aminooxy linkers bound to the carrier. The coupling reaction was carried out at a neutral pH and room temperature. The carrier protein was a non-toxic recombinant diphtheria toxin mutant. IgG antibody levels induced in young outbred mice by this new S. sonnei O-SPC conjugate were significantly higher then those elicited by the O-SP conjugates.

ELIGIBILITY:
* INCLUSION & EXCLUSION CRITERIA:

Healthy adults, 18 to 49 years of age of either sex who do not have any of the following conditions will be eligible to participate:

1. A chronic or progressive disease requiring chronic medication,
2. History of splenectomy or abnormal immune system,
3. History of neurological symptoms or signs, or mental illness,
4. Anaphylactic shock following administration of any vaccine or any other severe allergic reaction,
5. Women who are pregnant or intend to become pregnant during the vaccine study,
6. Had S. sonnei shigellosis in the past year or received a S. sonnei vaccine previously,
7. Have received systemic steroids during the month preceding Shigella vaccination,
8. Had cancer, HIV/AIDS, Hepatitis B or C, Guillain Barre Syndrome, chronic skin disease or have abnormal liver functions or blood counts.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-16; Primary Completion 2012-04-25 (Actual); Study Completion 2012-04-25 (Actual)

PRIMARY OUTCOMES:
Vaccine Safety

SECONDARY OUTCOMES:
Induction of IgG antibody type-specific immunity to shigellosis in adults.
Induction of higher levels of IgG antibody than with the previous experimental vaccines made with the full length O-SP

CONTACTS AND LOCATIONS:
Overall Officials: Germaine M Louis, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] Robbins JB, Kubler-Kielb J, Vinogradov E, Mocca C, Pozsgay V, Shiloach J, Schneerson R. Synthesis, characterization, and immunogenicity in mice of Shigella sonnei O-specific oligosaccharide-core-protein conjugates. Proc Natl Acad Sci U S A. 2009 May 12;106(19):7974-8. doi: 10.1073/pnas.0900891106. Epub 2009 Apr 3. PMID 19346477
- [Background] Taylor DN, Trofa AC, Sadoff J, Chu C, Bryla D, Shiloach J, Cohen D, Ashkenazi S, Lerman Y, Egan W, et al. Synthesis, characterization, and clinical evaluation of conjugate vaccines composed of the O-specific polysaccharides of Shigella dysenteriae type 1, Shigella flexneri type 2a, and Shigella sonnei (Plesiomonas shigelloides) bound to bacterial toxoids. Infect Immun. 1993 Sep;61(9):3678-87. doi: 10.1128/iai.61.9.3678-3687.1993. PMID 8359890
- [Background] Cohen D, Ashkenazi S, Green M, Lerman Y, Slepon R, Robin G, Orr N, Taylor DN, Sadoff JC, Chu C, Shiloach J, Schneerson R, Robbins JB. Safety and immunogenicity of investigational Shigella conjugate vaccines in Israeli volunteers. Infect Immun. 1996 Oct;64(10):4074-7. doi: 10.1128/iai.64.10.4074-4077.1996. PMID 8926071